CLINICAL TRIAL: NCT01060891
Title: Population Pharmacokinetic Study of Colistin in Patients Infected With Multiresistant Gram-negative Bacteria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Other Study IDs: COLI-POP
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Gram-negative Bacteria
Keywords: patients infected with with multiresistant gram-negative bacteria
MeSH Terms: interventions — Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: colimycin

SUMMARY:
Nosocomial infections have become a major health problem. They induced important use of antibiotics which is a preponderant factor for the development of bacterial resistance. The multi-resistance to antibiotics affects primarily Gram-negative bacteria. Some strains (as Acinetobacter or Pseudomonas) have become resistant to almost all antibiotics currently available, and the use of old molecules as Colistin may be the only alternative. However, there are few reliable data about Colistin and its PK characteristics. These data are essential to optimize its administration. The aim of the present study is to evaluate the pharmacokinetics of Colistin and its prodrug, colistimethate (CMS) after intravenous administration of Colistimethate alone or combined with inhaled Colistin in severely ill patients infected with multiresistant gram-negative bacteria

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 85 years
* Patients with nosocomial infection justifying Colistin.

Exclusion Criteria:

* Patients who received Colistin within 7 days prior to its inclusion, whatever the dosage or the route of administration
* Known hypersensitivity to Colistin or products of the polymyxin family
* Personal and family history for myasthenia
* Positive serology for HBV, HCV and HIV
* Positive pregnancy test or currently lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-05; Primary Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital - 2 rue de la Milétrie, Poitiers, France

REFERENCES:
- [Derived] Boisson M, Gregoire N, Cormier M, Gobin P, Marchand S, Couet W, Mimoz O. Pharmacokinetics of nebulized colistin methanesulfonate in critically ill patients. J Antimicrob Chemother. 2017 Sep 1;72(9):2607-2612. doi: 10.1093/jac/dkx167. PMID 28575278